CLINICAL TRIAL: NCT00840593
Title: A Prospective, Randomised 18 -Year Follow-up Study of Operative and Non-operative Treatment of Acute, Total Acromioclavicular Dislocation.
Brief Title: A Prospective, Randomised Long-term Follow-up of Operative Versus Non-operative Treatment of Gr. 3 Acromioclavicular Dislocation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Antti Joukainen, MD, PhD, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH5203037
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Acromioclavicular Joint; Dislocation; Surgical Procedures, Operative
Keywords: Acromioclavicular Joint; Dislocation; Trials, Randomized Clinical; Surgical Procedures, Operative
MeSH Terms: conditions — Joint Dislocations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Non-surgical group (Active Comparator): The non-surgical treatment consisted of immobilisation of the injured AC-joint in a Kenny-Howard-type splint for four weeks. The patient was encouraged in mobilisation of the elbow several times per day and the mobilisation of the shoulder with pendulum type movements were initiated four weeks after the injury. Active mobilisation of the shoulder was allowed six weeks after the injury.
  Interventions: Procedure: Non-surgical group
- 2 Surgical group (Active Comparator): The surgical treatment was accomplished within two days after the injury, and it consisted of an open reduction and fixation of the AC joint with two smooth Kirschner wires (2 mm in diameter) across the AC-joint. The K-wires were bent at the proximal ends, with suturing of the superior AC ligament. The position of Kirschner wires was confirmed during the operation using C-arm transillumination. The articular disc of AC joint was removed if it was damaged. Postoperative care consisted of immobilisation of the AC joint in a sling, (Polysling, body band) for four weeks and the mobilisation of the shoulder started four to six weeks later in a similar manner as in the non-operative group.
  Interventions: Procedure: Surgical group

INTERVENTIONS:
Procedure: Non-surgical group — The non-surgical treatment consisted of immobilisation of the injured AC-joint in a Kenny-Howard-type splint for four weeks. The patient was encouraged in mobilisation of the elbow several times per day and the mobilisation of the shoulder with pendulum type movements were initiated four weeks after the injury. Active mobilisation of the shoulder was allowed six weeks after the injury.
  Arms: 1. Non-surgical group
Procedure: Surgical group — The surgical treatment was accomplished within two days after the injury, and it consisted of an open reduction and fixation of the AC joint with two smooth Kirschner wires (2 mm in diameter) across the AC-joint. The K-wires were bent at the proximal ends, with suturing of the superior AC ligament. The position of Kirschner wires was confirmed during the operation using C-arm transillumination. The articular disc of AC joint was removed if it was damaged. Postoperative care consisted of immobilisation of the AC joint in a sling, (Polysling, body band) for four weeks and the mobilisation of the shoulder started four to six weeks later in a similar manner as in the non-operative group.
  Arms: 2 Surgical group

SUMMARY:
The purpose of this study is to compare the long-term clinical and radiological results of operative and conservative treatment of Tossy type 3 acromio-clavicular dislocation.

DETAILED DESCRIPTION:
The optimal treatment of Rockwood type 3 AC joint injuries is still controversial. This controversy results from the low level of evidence of the early literature and the evaluation of all AC joint injuries with a type I through III classification system.

There are no prospective randomized controlled long-term studies on the treatment of Tossy type 3 AC dislocation using primary repair and minimal pin fixation.

In this study, the non-surgical treatment consisted of immobilisation of the injured AC-joint in a Kenny-Howard-type splint for four weeks. The surgical treatment consisted of an open reduction and fixation of the AC joint with two smooth Kirschner wires (2 mm in diameter) across the AC-joint. The K-wires were bent at the proximal ends, with suturing of the superior AC ligament.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Tossy grade 3 AC-dislocation was recruited between the years 1989 and 1991 at Kuopio University Hospital for a randomized controlled study
* A written informed consent.

Exclusion Criteria:

* Not written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-02; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Presence of delayed surgical procedure to treat the AC joint dislocation pathology | from 18 to 20 years

SECONDARY OUTCOMES:
Grading of the AC dislocation using Rockwood classification (3-6) | 18-20 years
AC joint width in the middle of the joint (mm) | 18-20 years
Distance between proc. coracoideus and clavicle (coracoclavicular interspace) in Zanca projection, compared to non-injured side(mm) | 18-20 years
Osteolysis of clavicle (none, mild, moderate, severe) for follow-up radiographs | 18-20 years
Presence of calcification of CC ligaments (yes/no) | 18-20 years
Osteoarthrosis using modified Kellgren-Lawrence classification for follow-up radiographs | 18-20 years
Other pathologic condition of the shoulder (eg. osteoarthrosis of the glenohumeral joint, elevation of the humerus, calcific deposits of cuff) and the description of it | 18-20 years
The source (mechanism) of the AC dislocation injury (eg. falling, collision | 0 day
Patient age at the time of injury (years) | 0 day
Patient weight (kg) | 18 - 20 years
Patient length (cm) | 18 - 20 years
Occupation | 18 - 20 years
Grading of the work (light, heavy work, retired) | 18 - 20 years
Presence of other pathologic conditions or operative treatments for the shoulder, AC joint or other part of shoulder, description of it | 18 - 20 years
Larsen score | 18-20 years
Simple Shoulder Test (SST) | 18-20 years
UCLA score | 18-20 years
Constant score | 18-20 years
Oxford score | 18-20 years
Instability experiences of the AC joint (none, sometimes = less than 10 times a year, often = more than 10 times year) | 18-20 years
Pain (VAS, cm) related to instability experience of AC joint | 18-30 years
Range of motion of the shoulder (flexion, abduction, horizontal adduction, degrees | 18-20 years
Palpation of the AC joint (normal, prominent but stable, unstable) | 18-20 years
Pain of palpation (no or yes) | 18-20 years
Cross arm test (pain in AC joint, no/yes) | 18-20 years
Other pathologic findings of the shoulder in the clinical examination and the description of it | 18-20 years

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital, Kuopio, Kuopio, Finland